CLINICAL TRIAL: NCT04680104
Title: Prospective Observational Study Comparing Calcium and Sodium Levofolinate in Combination With 5FU/or in FOLFIRI Regimen
Brief Title: Prospective Observational Study Comparing Calcium and Sodium Levofolinate in Combination With 5-Fluorouracil (5FU) /or in FOLFIRI Regimen
Status: Completed | Type: Observational
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IRST159.01
Record Dates: First submitted 2020-12-15; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Gastrointestinal Cancer; CALCIUM LEVOFOLINATO (Ca-lev); SODIUM LEVOFOLINATO (Na-lev)
Keywords: Levofolinic Acid; Gastrointestinal Cancer; FOLFIRI
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Infusion of Na-Lev plus 5-FU (unique administration by one 48h-infusional pump)
- Cohort B: Infusion of Ca-Lev followed by infusion of 5-FU (two separated administrations by using one plastic bag followed by one 48h-infusional pump)

SUMMARY:
Prospective observational study comparing calcium and sodium levofolinate in combination with 5FU/or in FOLFIRI regimen on patients affected by gastrointestinal cancer (any site of disease along with gastrointestinal tract) who have been prescribed FOLFIRI in standard clinical practice.

DETAILED DESCRIPTION:
This is an observational, perspective trial on patients affected by gastrointestinal cancer (any site of disease along with gastrointestinal tract) who have been prescribed FOLFIRI in standard clinical practice. All patients will be treated and monitored according to the local clinical practice. No additional procedures/patient visits in comparison with the usual clinical practice are planned for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients affected by gastrointestinal cancer including:

   * advanced colon-rectal cancer,
   * biliary tract cancer,
   * pancreatic carcinoma,
   * advanced gastric or gastro-esophageal junction adenocarcinoma requiring treatment according to folfiri schedule
2. Participant is willing and able to give informed consent for participation in the study.
3. Male or Female aged >18 years.
4. Life expectancy > 3 months
5. Performance Status (PS) 0-1

Exclusion criteria:

1. Patients with known hypersensitivity to 5-FU or folinic acid , or to any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by gastrointestinal cancer requiring treatment according to FOLFIRI schedule
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 2 years
  Safety profiles of Na-Lev and Ca-Lev when administered in combination with 5-FU in FOLFIRI regimen to cancer patients under standard clinical practice. Reported Adverse Events (AE) will be summarized by system organ class, seriousness, severity (according to NCI -Common Terminology Criteria for Adverse Events, CTCAE version 4.0) and relationship to study drug. Comparison between groups will be performed using non parametric statistical test.

SECONDARY OUTCOMES:
organizational impact on Drug production | up to 2 years
  organizational impact that the introduction of Na-Lev would have on Drug production and delivery. The set-up times of preparation of Na-lev (by manual procedure) with respect to Ca-lev will be measured: for each individual therapy prescribed by clinicians the timing of the manual preparation in Official Pharmaceutical Lab (LFO) will be measured by chronometer, for the entire duration of each production line.
economical impact | up to 2 years
  economical impact hat the introduction of Na-Lev would have on Drug production and delivery. The set-up times of preparation of Na-lev (by manual procedure) with respect to Ca-lev will be measured: after preparation, the difference in waste of residual drug will be measured (if present) for each production. Quantity of residual drugs will be reported for each product line taking account of weight of enrolled patients.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Passardi, MD, Principal Investigator — Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Passardi A, Monti M, Donati C, Foca F, Pagan F, Rapposelli I, Ruscelli S, Bartolini G, Valgiusti M, Matteucci L, Sullo F, Sbaffi S, Crudi L, Frassineti GL, Masini C. Prospective Observational Study Comparing Calcium and Sodium Levofolinate in Combination with 5-Fluorouracil in the FOLFIRI Regimen. Oncologist. 2021 Aug;26(8):e1314-e1319. doi: 10.1002/onco.13762. Epub 2021 Apr 22. PMID 33764600